CLINICAL TRIAL: NCT01863797
Title: Trial on Early Induction Versus Expectant Management of Nulliparous Women With a Prolonged Latent Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Elena Bräne, RNM, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2007/65-31/2; 2007/65-31/2 (Other: EPN Stockholm)
Record Dates: First submitted 2013-05-20; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Nulliparous Women With Prolonged Latent Phase

ARMS (2):
- Early induction (Active Comparator): Induction was performed if membranes were still intact and cervical dilation was less than four centimetres five hours after medication for therapeutic rest. For participants with an unripe cervix intravaginal prostaglandin E2 (PgE2, dinoproston) was used. A transcervical catheter (BARD) was inserted if this procedure was possible 19 and if cervical dilatation permitted, amniotomy was performed. The physician in charge performed all assessments and procedures except amniotomy.
  When the participants reached the active phase they were monitored according to the clinical guidelines.
  Interventions: Other: Early induction
- expectant management (Experimental): The participants in the control group awaited spontaneous onset of labour as long as possible (expectant management). If contractions had ceased or subsided after the therapeutic rest women could be discharged from hospital, but were still included in the study. When reaching the active phase of labour women were monitored according to the clinical guidelines.
  Interventions: Other: Expectant mamagement

INTERVENTIONS:
Other: Early induction
  Arms: Early induction
Other: Expectant mamagement
  Arms: expectant management

SUMMARY:
The purpose of the study was to compare early induction versus expectant management regarding outcome and experience of delivery in nulliparous women with a prolonged latent phase.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy nulliparous women and normal pregnancies (in vitro-fertilisation included)
* with a singleton fetus in cephalic presentation,
* gestational age between 37+0 and 41+6,
* continuous contractions exceeding 18 hours impeding rest (women's report),
* a cervical dilation of less than four centimetres and intact membranes. Gestational age was confirmed by ultrasound in the first trimester.

Women had to be able to read, understand and speak Swedish.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome was mode of delivery (caesarean sections and vaginal deliveries (spontaneous and instrumental)) | Participants will be followed for the duration of hospital stay, an expected average of 3 days

SECONDARY OUTCOMES:
Maternal outcome measure included experience of delivery | Experience of delivery was assessed two days after delivery
  Wijma Delivery Experience Questionnaire - validated instrument. The 33 question questionnaire was filled in by the participance two days after delivery at postnatal care unit or at home.

OTHER OUTCOMES:
Maternal outcome measures included duration of labour, labour analgesia, intrapartum exogenous oxytocin stimulation, partum haemorrhage, number of sphincter tears. | Duration of labour, labour analgesia, intrapartum exogenous oxytocin stimulation were measured from cervical dilatation of 4 cm until delivery. Post partum hemorrhage was measured two hours after delivery. Sphincter tear measure directly after delivery.
  Duration of labour was measured in hours from cervical dilatation of four cm until delivery. Only the most active analgesia was recorded during active delivery (from cervical dilatation of four cm until delivery). Intrapartum exogenous oxytocin stimulation during active labour was recorded (yes or no). Post partum hemorrhage was measured from delivery and until two hours after delivery.
Neonatal outcomes; birth presentation, Apgar score below 7 and cord artery metabolic acidosis, admission to neonatal intensive care (NICU), birth weight and child's head circumference | Neonatal outcomes were measured from delivery and until two days after delivery.
  Birth presentation was assessed at delivery. Apgar score was assessed five minutes after delivery and cord artery metabolic acidosis assessed at delivery. Admission to NICU was measured from delivery and until two days after delivery. Birth weight and child's head circumference was measured in average two hours after delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Förlossningen, Danderyd Hospital, Stockholm, Stockholm County, Sweden